CLINICAL TRIAL: NCT05513885
Title: Bacterial Ecology of Pilonidal Cysts
Acronym: PILOBAC
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: COS-RGDS-2020-12-003
Record Dates: First submitted 2022-06-23; First posted 2022-08-24 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Pilonidal Cysts
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bacterial ecology of pilonidal cysts Single centre retrospective exploratory study of medical data contained in the medical records of patients operated on in the centre between 01/08/2020 and 30/11/2020.

DETAILED DESCRIPTION:
From the medical records of a series of patients treated for pilonidal cysts:

1. Describe the bacteriological analyses performed on a series of non-abscessed pilonidal cysts before laser treatment
2. Compare the bacterial flora of cysts operated on in the first instance and those reoperated on

This is a retrospective monocentric study of medical data contained in the medical records of patients operated on for pilonidal cysts and who received the same protocol:

* Antibiotic prophylaxis (injection of 2g of Augmentin)
* Treatment of the cyst by laser, under general anaesthesia, after dilatation of the pilonidal sinus, evisceration and bacteriological swabbing.
* Post-operative monitoring and local care

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older,
* Patient who has been informed about the research;
* Patient with a pilonidal cyst treated with Holmium Laser during a scheduled procedure.

Exclusion Criteria:

* Patient under legal protection, guardianship or curatorship;
* Patient who has indicated his opposition to the use of his data;
* Patient undergoing emergency surgery for an abscess.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients operated on for pilonidal cysts and who received the same protocol:
  * Antibiotic prophylaxis (injection of 2g of Augmentin)
  * Treatment of the cyst by laser, under general anaesthesia, after dilatation of the pilonidal sinus, evisceration and bacteriological swabbing.
  * Post-operative monitoring and local care
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Main germs incidence rate | Day 1
  Calculation of the the incidence rates of the main germs

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de la Sauvegarde, Lyon, France

IPD SHARING:
Plan to Share IPD: No